CLINICAL TRIAL: NCT05289869
Title: The HILIO Trial: High vs. Low Oxytocin Dosing for Induction of Labor in Pregnant Patients With Obesity- PILOT STUDY
Brief Title: A Pilot Study: High Versus Low Oxytocin Dosing for Induction of Labor in Pregnant Patients With Obesity
Acronym: HILIO-PILOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Heather Frey, MD, MSCI, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021H0432
Record Dates: First submitted 2022-02-25; First posted 2022-03-22 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pregnant Patients With Obesity
Keywords: Oxytocin; Pregnant patients with obesity; Induction of labor
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, research staff, and clinical care providers will be blinded to the dosing regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High-dose oxytocin regimen (Experimental): Starting dose 6 mU/min and increased by 6 mU/min every 30 minutes until adequate contractions achieved, at the discretion of the obstetric providers.
  Interventions: Drug: High-dose oxytocin
- Low-dose oxytocin regimen (Experimental): Starting dose 2 mU/min and increased by 2 mU/min every 30 minutes until adequate contractions achieved, at the discretion of the obstetric providers.
  Interventions: Drug: Low-dose oxytocin

INTERVENTIONS:
Drug: High-dose oxytocin — Starting dose 6 mU/min and increased by 6 mU/min every 30 minutes until adequate contractions achieved, at the discretion of the obstetric providers.
  Arms: High-dose oxytocin regimen
Drug: Low-dose oxytocin — Starting dose 2 mU/min and increased by 2 mU/min every 30 minutes until adequate contractions achieved, at the discretion of the obstetric providers.
  Arms: Low-dose oxytocin regimen

SUMMARY:
Pregnant patients with obesity are more likely to undergo induction of labor and have a higher risk of failed induction compared to patients with normal weight. The association between maternal obesity and labor dysfunction leading to cesarean delivery is poorly understood. Oxytocin is the mostly common medication used in induction of labor, yet optimal dosing of this medication is unknown. Studies have suggested that patients with obesity may be less responsive to oxytocin. This trial will compare a high and low dose oxytocin dosing regimen for the induction of labor in women with obesity.

DETAILED DESCRIPTION:
This study is a pragmatic single center randomized, double blinded controlled trial. Nulliparous women with a pre-pregnancy body mass index (BMI) ≥30 kg/m2 undergoing induction of labor at ≥37 weeks' gestation will be eligible for enrollment. Women will be randomly allocated to receive oxytocin using either a high-dose or low-dose regimen. Patients, providers, and research staff will be blinded to the dosing regimen. All other aspects of obstetric management will be at the discretion of the patient's clinical care team.

Postpartum maternal, neonatal, and delivery outcomes will be collected. Postpartum data through hospital discharge will be collected from the medical record. Information about complications following hospital discharge through 6 weeks after delivery will be collected during a research follow-up telephone call performed 6-8 weeks following delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparity
2. Maternal age >18 years
3. Gestational age ≥37w0d
4. Induction of labor, defined as initiation of labor with medication or intracervical Foley catheter in a patient without observed spontaneous cervical change and <6 contractions per hour (average of one contraction every 10 minutes) at the time of initial presentation. Women with prelabor rupture of membranes (PROM) can be included if the other criteria are also met with regards to cervical dilation and contractions.
5. Singleton gestation
6. Cephalic presentation
7. Indication for oxytocin use in the first stage of labor
8. No contraindication to labor or vaginal delivery
9. Pre-pregnancy BMI ≥30 kg/m2 based on patient report and confirmed by pre-pregnancy or first trimester weight as recorded in the medical record
10. Cervical dilation ≤4 cm at time of initiation of induction

Exclusion Criteria:

1. Fetal demise
2. Major fetal congenital malformation or known chromosomal abnormality
3. Prior uterine surgery (e.g., cesarean, myomectomy)
4. Non-reassuring fetal wellbeing as indication for induction
5. Intraamniotic infection suspected or diagnosed prior to randomization
6. Non-English
7. Multifetal gestation
8. Gestational age <37 weeks
9. Spontaneous labor
10. Cervical dilation > 4 cm at initiation of induction
11. Initiation of oxytocin in the second stage of labor
12. Use of oxytocin prior to randomization or planned use of oxytocin with foley catheter for cervical ripening
13. Fetal malpresentation
14. Estimated fetal weight >4500 g in a patient with diabetes, or estimated fetal weight >5000 g in a non-diabetic patient
15. Abnormal placentation (e.g. previa, suspected placenta accreta spectrum)
16. Physician/provider or patient refusal

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-dose Oxytocin Regimen | Low-dose Oxytocin Regimen
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High-dose: Group randomized to high-dose oxytocin regimen
- Low-dose: Group randomized to low-dose oxytocin regimen
- Total: Total of all reporting groups
Arm/Group | High-dose | Low-dose | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years]
  Maternal age | 25.5 (4.53) | 26.9 (6.06) | 26.2 (5.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic Black | 3 | 1 | 4
  Race/ethnicity: Non-Hispanic White | 7 | 7 | 14
  Race/ethnicity: Hispanic | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Delivery BMI, Continuous [Median (Inter-Quartile Range); unit: kg/m^2] | 41.8 [34.9 to 45.3] | 41.4 [35.1 to 45.1] | 41.6 [35.1 to 45.2]
Delivery BMI ≥40 [Count of Participants; unit: Participants] | 6 | 6 | 12
Gestational age, continuous [Median (Inter-Quartile Range); unit: weeks] | 38.0 [37.1 to 40.1] | 39.1 [38.0 to 40.1] | 38.7 [37.6 to 40.1]
Admission Bishop score <5 [Count of Participants; unit: Participants] | 8 | 7 | 15
Maximum oxytocin dose [Median (Full Range); unit: mu/min] | 16.5 [6 to 36] | 10 [2 to 26] | 13 [2 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Delivered by Cesarean
Time Frame: Until delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 3 | 3

2. Secondary Outcome: Duration of Time From Start of Induction to Delivery
Description: Time from start of induction with medication or Foley catheter until delivery
Time Frame: From start of induction to delivery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
hours | 22.6 [15.9 to 30.3] | 24.7 [21.2 to 34.7]

3. Secondary Outcome: Duration of the First Stage of Labor
Description: Time from start of labor to complete dilation
Time Frame: From start of induction to delivery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 8 | 7
hours | 17.3 [14.2 to 28.6] | 21.4 [16.3 to 26.6]

4. Secondary Outcome: Occurrence of Tachysystole
Description: Defined as more than 5 contractions in 10 minutes averaged over 30 minutes
Time Frame: From start of induction to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 5 | 3

5. Secondary Outcome: Incidence of Uterine Rupture
Description: Defined as a complete disruption of all uterine layers including serosa
Time Frame: From start of induction to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

6. Secondary Outcome: Incidence of Clinical Chorioamnionitis
Description: Defined based on clinical diagnosis as documented by the clinical care team
Time Frame: From start of induction thorough delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 3 | 1

7. Secondary Outcome: Incidence of Postpartum Maternal Infectious Morbidity
Description: Defined as a composite outcome of endomyometritis, puerperal sepsis, or surgical site infection as documented in the the clinical record
Time Frame: Within 6 weeks following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

8. Secondary Outcome: Incidence of Maternal Death
Time Frame: Within 6 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

9. Secondary Outcome: Incidence of Immediate Postpartum Hemorrhage
Description: Defined as >1000 mL of blood loss within 24 hours of delivery
Time Frame: Within 24 hours of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 0 | 1

10. Secondary Outcome: Incidence of Maternal Blood Transfusion
Description: Defined as need for blood transfusion
Time Frame: From randomization through hospital discharge up to 6 weeks portpartum
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 0 | 1

11. Secondary Outcome: Incidence of Maternal ICU Admission
Time Frame: From randomization through 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

12. Secondary Outcome: Incidence of Composite Neonatal Morbidity Outcomes
Description: Apgar score <5 at 5 min, arterial cord pH <7.0 or base deficit >12 mmol/dL, perinatal death
Time Frame: Within 6 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 1 | 1

13. Secondary Outcome: Incidence of NICU Admission
Time Frame: Within 6 weeks of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
Participants | 1 | 2

14. Secondary Outcome: Maternal Length of Stay
Description: Duration of hospitalization for delivery
Time Frame: Within 6 weeks of delivery
Measure: Median (Full Range); unit: days
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
days | 3 [2 to 5] | 3 [2 to 5]

15. Secondary Outcome: Neonatal Length of Stay
Description: Duration of birth hospitalization
Time Frame: Within 6 weeks of delivery
Measure: Median (Full Range); unit: days
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 10
days | 2 [1 to 3] | 2 [2 to 6]

16. Secondary Outcome: Perception of the Labor, Birth, and Postpartum Experience
Description: Patient perception as measured using the validated Childbirth Perception Scale. This is a 12-item instrument developed to assess a patient's perception of the labor and delivery experience. Each item is formatted on a four-point scale ranging from 0 to 3. The overall range in total score is 1-36 with higher scores indicating a less positive perception.
Time Frame: Assessed within 12-96 hours after delivery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 10 | 9
score on a scale | 14 [9 to 16] | 9 [7 to 14]

17. Secondary Outcome: Labor Agentry Score
Description: Patient perception of labor agentry as measured using validated Labor Agentry Scale. This 29-item tool was developed to assess a patient's expectancies and experiences with control in labor. Each item is scored 1 to 7. Overall total score can range from 29-201 with higher scores indicated greater perceived control during childbirth.
Time Frame: Assessed within 12-96 hours after delivery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | High-dose | Low-dose
Number analyzed (Participants) | 8 | 9
score on a scale | 139.5 [138 to 174] | 185 [169 to 190]

ADVERSE EVENTS:
Time Frame: 6 weeks following delivery
Description: An adverse event (AE) will be defined as any untoward or unfavorable medical occurrence in a study participant, whether or not considered related to the subject's participation in the research.
Arm/Group | High-dose | Low-dose
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-dose (N=10) | Low-dose (N=10)
Hospital readmission (Investigations) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT05289869/Prot_SAP_000.pdf